CLINICAL TRIAL: NCT03161197
Title: Pain Relief Intervention of Meditation in Renal Disease
Brief Title: Pain Relief Intervention of Meditation in Renal Disease (PRIMER)
Acronym: PRIMER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1503016044
Record Dates: First submitted 2017-05-04; First posted 2017-05-19 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Chronic Kidney Diseases; Renal Disease; Chronic Kidney Failure; End Stage Renal Disease
Keywords: CKD, Dialysis, ESRD; Mindfulness-Based Stress Reduction (MBSR)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Kidney Failure, Chronic | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Dialysis patients will receive the intervention individually while on dialysis. Dialysis is an optimal time for conducting interventions as patients are there for 3-4 hours every 3 days. For 8-10 weeks (which will begin the week after the baseline interview). Chronic Kidney Disease (CKD) patients will receive the intervention in group setting. Since CKD patients only come to see their nephrologist once a month, all CKD potential participants will be invited to attend eight consecutive weekly sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention consists of 8-10 sessions consisting of mindfulness-based stress reduction. Key components of what the intervention consists relate to stress management, breathing, and meditation exercises, as well as, techniques aimed at improving relations with others, sense of mastery and purpose in life. Additionally, during every point of contact subjects will be asked how often they utilized the strategies they were taught. This information will be helpful in understanding each subject's individual level of mastery and proficiency in Mindfulness-Based Stress Reduction (MBSR).
  Interventions: Behavioral: Mindfulness-Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — The intervention consists of mindfulness-based stress reduction. Key components of what the intervention consists relate to stress management, breathing, and meditation, as well as, techniques aimed at improving relations with others, sense of mastery and purpose in life. Additionally, the intervention subjects, during every point of contact, will be asked how often they utilized the strategies they were taught. This information will be helpful in understanding each subject's individual level of mastery and proficiency in Mindfulness-Based Stress Reduction (MBSR).
  Other Names: MBSR

SUMMARY:
Kidney Disease subjects will be recruited to take part of a mindfulness-based stress reduction intervention for 8-10 sessions. All subjects will complete a baseline interview, one follow-up at 3 months and the close out interview at 5 months.

DETAILED DESCRIPTION:
Kidney Disease subjects will be recruited from multiple locations within the Rogosin Institute Dialysis Center to take part of a mindfulness-based stress reduction intervention. The intervention consists of meet with a researcher and/or research assistant on a weekly basis. Dialysis patients will receive the intervention individually while on dialysis. Dialysis is an optimal time for conducting interventions as patients are there for 3-4 hours every 3 days. For 8-10 weeks (which will begin the week after the baseline interview). Chronic Kidney Disease (CKD) patients will receive the intervention in group setting. Key components of what the intervention consists relate to stress management, breathing, and meditation exercises, as well as, techniques aimed at improving relations with others, sense of mastery and purpose in life. Additionally, during every point of contact, will be asked how often they utilized the strategies they were taught. This information will be helpful in understanding each person's individual level of mastery and proficiency in Mindfulness-Based Stress Reduction (MBSR). All subjects will complete a baseline interview, one follow-up at 3 months and the close out interview at 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Kidney Disease (CKD) and ESRD on dialysis for over 6 months and who are willing to consent. English speakers only, 18 years of age or older

Exclusion Criteria:

* Patients with severe cognitive or psychiatric impairment will be excluded. Patients who are not willing to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in Pain: Participants self-report | 6 months
  Participants self-report

CONTACTS AND LOCATIONS:
Overall Officials: Carla Boutin-Foster, MD, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- See also: The Translational Research Institute for Pain in Later Life (TRIPLL) is an NIA funded Edward R. Roybal center with a focus on chronic pain — http://tripll.org/